# Assessing the Feasibility of Economic Approaches to Prevent Substance Abuse Among Adolescents

NCT Number: NCT05597865

**Study Protocol** 

Approved: 03 November 2022

# Assessing the Feasibility of Economic Approaches to Prevention of Substance Abuse among Adolescents

| Table of Contents<br>SPECIFIC AIMS | 2 |
|--------------------------------------------------------|----|
| Study objectives | |
| RESEARCH STRATEGY | |
| A.1. SIGNIFICANCE. | 3 |
| A.2. THEORETICAL FRAMEWORK. | |
| B. INNOVATION. | 4 |
| C. APPROACH | 5 |
| C.1. Study Team | 5 |
| C.2. Research design and study sites | 6 |
| C.3. Inclusion criteria. | |
| Exclusion criteria | 6 |
| C.4. Recruitment of participants and informed consent. | 7 |
| C.5. Data collection and assessment | 7 |
| C.6. Description of the RCT. | 7 |
| C.7.1 Quantitative Data analysis. | 8 |
| C.7.2. Qualitative data analysis | 9 |
| C.7.3. Data integration. | 9 |
| C.8. Potential challenges and alternative strategies | 9 |
| C.9. Dissemination. | 9 |
| D. TIMELINE. | 9 |
| E DEFEDENCES | 10 |



#### SPECIFIC AIMS

Adolescent alcohol and drug use (ADU) is a growing public health concern globally, especially in low resource settings such as Sub-Saharan Africa (SSA), where the epidemics of ADU and HIV/AIDS are co-occurring. ADU plays a significant role in the epidemiology of HIV among adolescents and young adults in SSA, who accounted for over 40% of new infections globally in 2019.¹ ADU is associated with higher rates of HIV risk behaviors such as condomless sex,² and lower rates of HIV testing.³-5 Among adolescents and youth living with HIV (AYLHIV), ADU is a significant barrier to achieving positive HIV treatment outcomes including enrollment and retention in HIV care, 6 adherence to antiretroviral therapy, 7-9 and achieving viral suppression. 8,10 Among HIV-infected adults, it has been shown that alcohol and drug misuse increase AIDS mortality, even among virally suppressed and medication adherent persons. 11-13 Uganda, one of the poorest countries in SSA, has high rates of HIV/AIDS (6.2%) 14 and alcohol use, 15 and illicit drug use is on the increase. 16 Previous studies have reported high rates of alcohol consumption among adults living with HIV. 17-19 Fishing communities – a key vulnerable population in Uganda<sup>20</sup> - have high levels of ADU including among adolescents and youth, 16,21-23 which lead to poor HIV prevention and care outcomes.

ADU typically onsets in adolescence as an experimental behavior that may escalate into problematic use and disorders. <sup>24,25</sup> In addition to mental health problems, <sup>26</sup> poverty, <sup>27-29</sup> poor parental supervision, <sup>30</sup> community norms related to drug use, <sup>31,32</sup> and developmental risk factors such as risk-taking, social roles and social transitions influence risk for ADU. <sup>33-35</sup> AYLHIV in particular experience numerous stressors (e.g. bereavement, HIV stigma and discrimination, death, worry, and chronic pain) <sup>36-38</sup> and mental health problems (e.g. depression and hopelessness), <sup>39-42</sup> which increase their risk for ADU. Consistent with motivational theories of alcohol and drug use, <sup>43-47</sup> AYLHIV may use alcohol and drugs as a mechanism for coping with stress and mental health problems such as depression, <sup>45,48,49</sup> which are common among AYLHIV. Household poverty, which is rampant in AIDS-affected households, <sup>50</sup> is associated with an increased risk for ADU. Despite our knowledge of the higher risk for ADU among AYLHIV, <sup>52-55</sup> there is lack of evidence-based interventions targeting ADU risk among AYLHIV.

Efforts to prevent ADU are rooted predominantly in the substance use risk reduction/protection enhancement model<sup>56</sup> and require understanding of the risk and resilience factors for ADU. Only 10 ADU interventions have been evaluated in SSA: most have been ineffective in preventing or reducing ADU and none of these interventions has targeted AYLHIV. The majority of these interventions, which are largely school-based, focus on individual and intra-personal risk factors for ADU, without attention to structural risk/resilience factors for ADU. The few existing studies on ADU among AYLHIV have been conducted in high-income countries. These studies focus on younger adolescents yet ADU typically emerges and escalates in middle-late adolescence. Further, these studies rely on self-reports of ADU which can be undermined by under-reporting of ADU. To address these challenges, we propose a study titled *Assessing the Feasibility of Economic Approaches to Prevention of Substance Abuse among Adolescents*. The study will investigate the epidemiology, underlying risk and resilience factors for ADU among AYLHIV and evaluate the effects of a economic empowerment intervention on ADU among AYLHIV. We propose to utilize biological measures of ADU to overcome challenges associated with self-reported ADU.

# Study objectives

The proposed study will investigate the following specific aims:

Aim 1a. Examine the prevalence and consequences of ADU in a cohort of 200 AYLHIV (ages 18-24) seen at six (6) HIV clinics in southwestern Uganda. We will utilize adolescent self-reports and biological measures of alcohol and drug use (urine).

<u>Aim 1b</u>. Using a mixed methods approach, identify the multi-level (individual, interpersonal, community and structural) factors associated with ADU among AYLHIV

<u>Aim 2</u>: Using a subset of the sample, explore the feasibility and short-term effects of a economic empowerment intervention on ADU among AYLHIV.

Our long-term goal is to better understand the epidemiology and consequences of ADU among AYLHIV in highrisk environments and evaluate a culturally tailored intervention that could prevent harmful ADU and improve the overall and long-term health and well-being of AYLHIV. The proposed study will be conducted in fishing communities located in three districts of the greater Masaka region of southwestern Uganda - a region heavily affected by HIV (12% prevalence vs national average of 6.2%) and high rates of household poverty and



alcohol/drug use. The findings from this proposed study will contribute to our understanding of the epidemiology, risk and resilience factors and consequences of alcohol and drug use among AYLHIV, in order to inform the development of effective ADU prevention intervention. If warranted, these findings will inform the design of an R01 grant to examine the long-term effects of a family-based economic empowerment intervention on ADU among AYLHIV.

#### RESEARCH STRATEGY

#### A.1. SIGNIFICANCE.

Adolescent alcohol and drug use (ADU) is a significant public health challenge in SSA. About 41.6% of adolescents in SSA have used at least one psychoactive agent.<sup>57</sup> Alcohol is the most commonly used drug;<sup>57</sup> one third of adolescents have used alcohol in their lifetime<sup>57,58</sup>, 22.5 million are current drinkers, and over 50% engage in heavy episodic drinking. 58 Alcohol use nearly doubles during the transition to adulthood, from 21.4% of adolescents aged 16-19 to 34.1% of young adults aged 20-24 years. 58 Uganda, one of the poorest countries in SSA, has the second highest rate of per capita alcohol consumption in SSA (15.1 liters of pure alcohol vs regional average of 6.2 liters of pure alcohol).15 Over 30% of Ugandan adolescents and youth have used alcohol<sup>59,60</sup> and about 20% misuse alcohol.<sup>16</sup> These estimates reach even greater magnitudes in the country's fishing villages - a key HIV vulnerable population- where ADU is normative. 61-64 A few studies have assessed ADU among AYLHIV. A study conducted in Rwanda found that 61% of AYLHIV receiving medication from a clinic had drunk alcohol within 6 hours prior to having sex.<sup>54</sup> In South Africa, a prior study found that 53.8% of the male AYLHIV and 5% of female AYLHIV had ever used drugs. 65,66 In Uganda, a recent cross-sectional study of 479 adolescents aged 12 - 17 years found that 5.9% reported use of at least one psychoactive substance, including alcohol (4.3%), marijuana (2.1%) and other drugs (2.1%) such as cocaine, glue and heroine. 67 ADU is a key driver of new HIV infections and poor HIV care outcomes in SSA. It is associated with HIV risk behaviors such as increased sexual risk-taking, 33,34,68 unprotected sex,2 early sexual debut,69-71 an increased number of sexual partners, 2,69,70 resulting in transmission of HIV.9,68,72,73 ADU is also associated with sub-optimal mental health e.g. depression<sup>74-76</sup> and suicidal ideation.<sup>77</sup> Among AYLHIV, ADU impedes adherence to anti-retroviral therapy (ART),<sup>7-9</sup> retention in care,<sup>6</sup> and viral suppression.<sup>8,10</sup> Among HIV-infected adults, ADU have been shown to increase susceptibility to AIDS mortality, even among HIV virally suppressed and medication adherent persons.11-13

AYLHIV are more vulnerable to ADU, which may affect their HIV care outcomes. Adolescence is a period characterized by exploration of new roles, identities, and behaviors including experimentation with ADU.78 A multitude of factors influence ADU and these include individual factors (e.g. sensation seeking, impulsivity, mental health), 79-84 interpersonal factors (e.g. peer pressure, parental drug use, poor parental monitoring) 85-95 and structural factors (e.g. availability of alcohol and drugs, exposure to ADU marketing, community drug use attitudes, laws and policies).85,90 AYLHIV, also experiment with ADU, which may escalate into problematic ADU. AYLHIV face numerous HIV-related psychosocial challenges including HIV stigma, bereavement, chronic pain, relationship stress and poverty, which heighten their risk for ADU. 96-98 Indeed, research reports indicate a higher burden of mental health problems among AYLHIV, 97,99-102 which may lead to ADU. The co-occurrence of mental health problems and ADU is common, including among AYLHIV. 103-110 Both ADU and mental health difficulties are associated with non-adherence to ART<sup>100,111-113</sup> and risky sexual behaviors among AYLHIV, 112,114-116 which could lead to secondary transmission of HIV and ART resistance due to non-adherence. 117-119 Poor mental health and poverty, which are rampant in poor countries, are significant risk factors for ADU. Poor mental health 106,120,121 and poverty<sup>27-29</sup> are rampant among HIV-affected households, and both are significant risks factor for acquiring HIV122 and for poor HIV treatment outcomes. 123,124 AYLHIV living in poverty-stricken households face greater challenges in accessing and sustaining HIV treatment due to economic factors such as lack of transport to clinics<sup>125,126</sup> and inadequate meals to support medication adherence, <sup>127-129</sup> which could lead to psychological distress and consequently, ADU. 130 Poverty adversely affects the quality of family relationships including parentchild communication, involvement<sup>131-133</sup> and parenting skills, <sup>134,135</sup> which increases susceptibility to emotional and behavioral challenges and increased risk for ADU. 93,95,132,136-140

**Evidence-based culturally tailored interventions to prevent ADU in AYLHIV are lacking**. Several studies have examined the risk and resilience factors for ADU<sup>56</sup> but few interventions targeting ADU have been tested in SSA. Only 10 ADU interventions have been evaluated in SSA<sup>79,141-149</sup> and only a few have been successful.<sup>79,142,143,146,148,149</sup> The majority have been implemented in school settings,<sup>79,145-149</sup> which may exclude adolescents in fishing communities that have high rates of school dropout. These interventions largely target

individual and interpersonal risk factors for ADU, with a focus on providing participants with information on ADU and its consequences, or building life skills. Only one intervention targeted the family<sup>144</sup> – an important developmental context for adolescents- with a focus on enhancing parenting skills. None of these interventions has targeted risk factors such as poverty and mental health that may undermine AYLHIV's coping skills and resources. Family-based economic empowerment (FEE) interventions have the potential to prevent ADU among AYLHIV by reducing poverty and its associated mental impacts, and also bolster AYLHIV and their families' resources to overcome the challenges associated with HIV. In our previous studies, we have utilized FEE strategies to reduce poverty, improve mental health and HIV care outcomes (e.g. medication adherence) among AYLHIV and other AIDS-affected adolescents in Uganda. 123,132,150-153 In this application, we propose to build on this growing evidence by examining the feasibility of utilizing FEE to address ADU among AYLHIV.

A.2. THEORETICAL FRAMEWORK. Our conceptual approach is informed by the socio-ecological model (SEM), 154 social causation and drift theories, 155 and asset theory. 156, 157 We have applied the SEM as a basis for investigating the contextually relevant risk and resilience factors for ADU. SEM posits that environmental factors fall into four broad domains: micro-, meso-, exo-, and macro systems and interactions within and between these domains determine behavior. This model has demonstrated effectiveness in identifying risk and resilience factors for prevention planning and intervention for ADU. 158-162 Social causation and social drift theories suggests that problem alcohol drinking may be both a response to and driver of poverty. 163 Acute and chronic stress associated with living in a poverty-impacted environment increases the likelihood of ADU, which causes further material/economic deprivation, hence fueling the cycle of alcohol misuse, and contributing to downward social mobility. Research in Uganda has reported a higher burden of alcohol and drug abuse among poor populations, 164 and many poverty-impacted Ugandan households engage in informal alcohol production for income-generating purposes.165 Impoverished youths are burdened with hopelessness due to lack of opportunities for improvement in their economic wellbeing. 166,167 As a result, for impoverished AYLHIV, they may be inclined to spend on instant pleasures such as alcohol and drugs as a coping mechanism since they are less likely to believe they can afford the costs associated with accessing and maintaining long-term care for HIV. Our proposed FEE intervention is based on Asset theory 168 and is intended to improve economic wellbeing and relieve poverty and its related consequences such as poor mental health, 169,170 and create a more hopeful/optimistic outlook for the future, thus reducing AYLHIV's engagement in risk-taking behaviors including alcohol and drug use. The proposed FEE will be one of the first studies to primarily examine the impact of FEE interventions on reducing ADU among AYLHIV in poverty-impacted communities.

# B. INNOVATION.

The proposed study innovates in the following ways: (1) We focus on older adolescents and young adults in a high-risk environment to elucidate the contextually relevant risk and resilience factors for ADU. Late adolescence and early adulthood are also when depression and other common mental health problems first emerge<sup>24,25</sup> yet majority of prior studies typically focus on younger adolescents. Most of the prior studies are constrained by the small samples of AYLHIV who report ADU. In this proposal, we focus on AYLHIV in fishing communities - vulnerable communities that have high rates of HIV and drug use. Together, this approach will ensure that we have a large sample size of AYLHIV reporting ADU, to explore the risk and resilience factors and their potential interactions. Such knowledge is necessary to develop effective interventions to prevent/reduce ADU among AYLHIV. (2) Our intervention targets the most commonly occurring risk factors for ADU (i.e. poverty and mental health problems). Only a few ADU interventions evaluated in SSA have targeted the family context. 144 No study has targeted poverty and its attendant impacts (e.g. mental health) as a risk factor for ADU. In this proposal, we will examine the feasibility, acceptability and short-term effects of a family-based economic empowerment intervention to reduce/prevent risky and hazardous alcohol drinking and drug use. The proposed FEE intervention is based on Asset theory 168 and is intended to improve economic wellbeing and create a more hopeful/optimistic outlook for the future, and thus reduce AYLHIV's engagement in risk-taking behaviors including alcohol and drug use. This will be one of the first studies to examine the impact of FEE interventions on reducing alcohol/drug use among AYLHIV in poverty-impacted communities. (3) We utilize biological measures to address limitations of self-reported drug use. Self-reported measures are frequently used to assess ADU yet, due to a number of factors including the legal drinking age, gender, religious practices, social/cultural acceptability around alcohol use, recall and social desirability bias, these measures result in significant under-reporting of ADU. 171,172 In addition, in SSA including Uganda, a substantial proportion of all alcohol consumed (~40% in LMICs and ~89% in Uganda<sup>173</sup>) is homemade,<sup>58</sup> which makes it difficult to determine the quantity of alcohol consumed. Hence, the inclusion of biological measures for ADU (urine test) can overcome



the measurement limitations encountered from the reliance on self-reported data to provide more accurate data on the prevalence of ADU.

#### C. APPROACH.

### C.1. Study Team.

We are a multidisciplinary team of investigators with expertise on AYLHIV's mental health, substance use and economic empowerment interventions. The team is co-led by Dr. Brathwaite (Lead MPI-Washington University in St. Louis-WUSTL) and Dr. Mutumba (MPI-University of Michigan). Dr. Brathwaite is a Research Assistant Professor WUSTL with training in Epidemiology and Population Health. She has research experience in substance use disorders and mental health among vulnerable/marginalized populations. She has published research focused on developing tools designed to predict future depression among adolescents in low and middle income countries, 174,175 and to predict depression and hopelessness among AYLHIV in Uganda. 176 She has experience working with vulnerable populations who use substances and has conducted research on substance use including persons who inject drugs in the UK, 1777-180 smoking among migrants from SSA and ethnic minority groups in Europe, 181-183 and research on the burden of alcohol use among households in Trinidad and Tobago. 184,185 More recently she has been involved in intervention research and analysis focused on the effects of schools-based mental health interventions and the impact of family-based economic empowerment interventions on adherence, economic and educational outcomes among AYLHIV in low resource communities in Uganda. Dr. Mutumba is an Assistant Professor at the University of Michigan with extensive experience conducting research among AYLHIV in Uganda. She has worked on several HIV clinical trials (UARTO187 and ARROW<sup>188</sup>), managed complex national studies in SSA, <sup>189,190</sup> and has extensive clinical and research experience working on adolescent substance use and mental health among AYLHIV across a range of settings. 36,191-196 Currently, she is collaborating with Dr. Ssewamala (Co-I) to test a multi-level school and familybased stigma reduction intervention that includes a family-based economic empowerment component for AYLHIV. Drs. Brathwaite and Mutumba have an established working relationship through their joint mentor and Co-I, Dr. Ssewamala who is also executive director of the International Center for Child Health and Development (ICHAD). Drs. Mutumba and Brathwaite will co-lead and oversee all aspects of the study including recruiting and training research assistants, developing of quantitative and qualitative data collection tools and study protocols, designing intervention materials, analyzing data, and disseminating findings. Dr. Brathwaite will be responsible to communicating with NIH. Dr. Filiatreau (Co-I) is a Postdoctoral Research Associate at WUSTL with training in Epidemiology and Public Health, and has research experience with AYLHIV in SSA. Her research centers on characterizing the psychosocial well-being of people living with HIV in resource-constrained settings and estimating the effects of mental health and ADU on HIV treatment and care in these populations. 197-202 More recently she has been involved in work using novel epidemiologic methods to estimate longitudinal HIV care continuum outcomes among people entering HIV care and quantify the effects of a range of both hypothetical and implemented interventions on these outcomes.<sup>203</sup> Dr. Filiatreau will assist Dr. Brathwaite in developing the quantitative survey instrument and support analysis of quantitative data, Dr. Ssewamala (Co-I), a Professor at WUSTL, is an accomplished expert in designing and implementing economic empowerment interventions and conducting research among AYLWHIV in Uganda. He has led multiple NIH-funded studies conducted in Uganda for the last 15+ years (Suubi, R21MH076475; Suubi-Maka, R34MH081763, Bridges, R01HD070727; Suubi+Adherence, R01HD074949). 131,151,204-211 These studies, all conducted in Uganda, have been highly acceptable and feasible, yielding positive health and development outcomes, and have had high adherence to study protocols. Dr. Ssewamala directs the International Center for Child Health and Development (ICHAD), which has an office with >50 full-time staff in the study region (see Resources). The proposed study will leverage the community connections established through these NIH-funded studies. Dr. Ssewamala is the mentor of Drs. Mutumba, Brathwaite and Filiatreau and will contribute to the designing and implementation of the economic empowerment intervention component of the study. Dr. Mugisha, Consultant is a clinical psychologist and Senior Lecturer of Mental Health at Kyambogo University in Uganda. He has worked extensively on mental health among varied populations including AYLHIV in Uganda. A skilled qualitative methodologist, he will contribute to developing qualitative interview guides, analysis and interpretation of study findings, and support Dr. Mwebembezi with study implementation. Dr. Mwebembezi (In-country PI) is the executive director of Reach-the-Youth (RTY), our local implementing partner in Uganda. His responsibilities will include: 1) recruiting, hiring and training research assistants to conduct cross-sectional and qualitative interviews; 2) ensuring staff have the necessary precertification including CITI Human Subjects Protection Training; 3) ensure all research activities are conducted per the approved research protocol.

# C.2. Research design and study sites.

We propose a mixed-methods study comprising 4 components: (1) focus group discussions (FGDs) with AYLHIV (n=20) and in-depth qualitative interviews (QI) with health providers (n=10). AYLHIV will be recruited from two randomly selected clinics; 10 participants per FGD; (2) a cross-sectional survey (CS) with 200 AYLHIV; (3) a



randomized control trial (RCT) with a sub-group of AYLHIV (n=100); and (4) two post-intervention FGD with AYLHIV (n=10 per study group). The study will be conducted in six

randomly selected HIV clinics located in fishing districts within the Greater Masaka region of Southwestern Uganda- a region heavily affected by HIV (12% prevalence vs. 6.2% national average)<sup>212</sup> with high rates of household poverty and alcohol use.<sup>62,213</sup> Urine tests for ADU will be conducted among all 200 AYLHIV who participate in the cross-sectional survey and among the 100 who participate in the RCT at the two time points. However, given the minimum and maximum detection times for different drugs of abuse in the urine, we will not exclude those with a positive self-report but negative urine test results from being included in the RCT. Additional analyses will explore the association between self-reported use and biomarkers.

#### C.3. Inclusion criteria.

The target populations for this study are: 1) AYLHIV, 2) healthcare providers at the selected HIV clinics. All study participants will be recruited from the selected HIV clinics. Inclusion criteria for clinics: 1) located in the - fishing districts with known HIV hotspots (i.e. 2 randomly selected clinics per district); 2) accredited by the Uganda Ministry of Health as a provider of ART; 3) currently have established services for AYLHIV. Inclusion criteria for AYLHIV: 1) male or female AYLHIV aged 18-24 years 2) medically diagnosed with HIV and aware of their HIV status; 3) enrolled in care at one of the selected HIV clinics. Inclusion criteria for health providers: health providers (1 - 2 per clinic) will be recruited from each of the selected clinics. Inclusion criteria for participants of the RCT: a sub-sample of AYLHIV (n=100) with a positive self-report for ADU will be randomly selected and randomly assigned at the clinic level (3 clinics per group) to either an intervention group (n=50) or a control group (n=50). AYLHIV from the control (n=10) and intervention groups (n=10) will participate in two FGDs at the end of the intervention.

**Exclusion criteria** for RCT and post-intervention FGD: any AYLHIV with negative self-report for ADU. **Exclusion criteria for all participants:** anyone with a significant cognitive impairment that interferes with their understanding of the informed consent process, or who is unable/unwilling to consent.

| SOCIO-ECOLO | GICAL FRAMEWORK | Time collected |
|---|---|---|
| Level | Risk/protective factor | |
| Individual | Socio-demographic: Gender; Age; orphanhood; education, income and unemployment; food insecurity <sup>214</sup> ; experienced homelessness; refugee; day/boarding school; urban/rural residence. <b>Mental health:</b> Depression, <sup>215</sup> hopelessness, <sup>216</sup> Optimism <sup>217</sup> ; Stress, <sup>218</sup> pain, <sup>219</sup> history of substance abuse <sup>220</sup> | CS, QI, FGD, RCT |
| Interpersonal/<br>Relationship | Loneliness <sup>221</sup> ; number of close friends; bullying; interpersonal violence; <sup>222,223</sup> social support <sup>224</sup> ; family cohesion <sup>225,226</sup> ; childhood abuse/trauma; family history of substance abuse, <sup>220</sup> sexual risk-taking <sup>228</sup> | |
| Community | Community norms; access to alcohol and illegal drugs | |
| Society | Educational campaigns; price and supply of alcohol, social stigma <sup>229</sup> | |
| Biomarkers | Urine alcohol and drug test | CS, RCT |
| Savings<br>deposits | Savings | Monthly ban statements |
| Assessments | Self-reported alcohol and drug use <sup>220</sup> ; Viral load from clinic records; Self-reported adherence <sup>230</sup> ; depressive symptoms <sup>215</sup> ; hopelessness <sup>216</sup> ; physical health conditions; sexual risk-taking <sup>228</sup> | RCT |



# C.4. Recruitment of participants and informed consent.

Recruitment strategies will build on RTY (local implementing partner) and ICHAD's long-standing relationships (>15 years) with 39 health clinics in the greater Masaka region. We will capitalize on recruitment procedures tested in previous SUUBI studies that involve collaborating with health clinics in the region (namely Suubi+Adherence: 1R01HD074949-01, Suubi+Adherence-R2: R01HD074949-07, and Suubi4Stigma: R21MH121141). All participants will be recruited from the selected HIV clinics. For the cross-sectional survey, 200 AYLHIV will be recruited from across six clinics located in the greater Masaka region. . The designated study contact at each health clinic will present the project to all eligible AYLHIV 18-24 years during their clinic visits. If there is interest, they will provide verbal consent to be contacted by the research study team. The study coordinator will contact interested AYLHIV to inform them about, the required extent of participation, the risks and benefits of participating, and to ask any questions. Written informed consent will be obtained from AYLHIV 18-24 years and from healthcare providers >18 years to participate. The written consent documents will emphasize the following elements: 1) participation in the study is voluntary; 2) responses to study questions are confidential; 3) participants can terminate their participation at any time and their decision to withdraw from the study will not affect their access to services they are currently receiving in any way; 4) participants may be contacted to participate in the RCT if eligible. A screening tool will be developed to assess whether participants meet the study inclusion criteria. Participants' data will be protected by a Certificate of Confidentiality, which protects the privacy of research subjects by prohibiting disclosure of identifiable, sensitive research information to individuals not involved in the research unless the participant consents.

#### C.5. Data collection and assessment.

After pilot testing of data collection interview tools, two separate <u>FGDs</u> will be conducted with AYLHIV (n=20) and in-depth <u>QIs</u> will be conducted with health providers (n=10). AYLHIV will be recruited from two randomly selected clinics; 10 participants per FGD. The FGDs and QIs will explore participants' perceptions on the multilevel risk and resilience factors associated with alcohol and drug use and recommendations for culturally appropriate ADU interventions for AYLHIV. Data from the qualitative phase will inform the questions to be asked in the cross-sectional survey. For the <u>cross-sectional survey</u>, 200 AYLHIV will complete an interviewer-administered survey comprising questions assessing their alcohol/drug consumption patterns and frequency as well as exposure to multi-level (individual, interpersonal, community and societal) factors that may be associated with risky and hazardous drinking and drug use among AYLHIV. To reduce social desirability bias, questions on ADU will be self-administered using audio computer assisted interviewing (ACASI). We refer to the social ecological framework<sup>231</sup> to guide data collection on the multiple levels of influence that are associated with harmful alcohol/drug use among AYLHIV (See Table 1 for socio-ecological framework and additional measures that will be collected at each time point). Questions assessing the presence of common mental disorders and the presence of other physical health conditions will be included.

<u>Biological measures:</u> A trained study research assistant will collect and test a urine specimen from each participant. The urine sample will be tested for up to 16 classes of the most commonly abused illicit drugs using the T-Cup 16 panel Compact Instant Drug Test Cup at the study site. The T-Cup can detect alcohol in the urine from as early as 8 hours to up to 80 hours after consumption. Minimum and maximum detection times for illicit drugs of abuse range from one hour to 40 days depending on the drug. AYLHIV will be tested during the cross-sectional survey and at baseline and 6-months follow-up during the RCT.

#### C.6. Description of the RCT.

For the RCT, 100 AYLHIV with a positive self-report or urine ADU test (based on data from the cross-sectional survey) will be randomly recruited from the six clinics and randomly assigned at the clinic level (3 clinics per group) to either the control (n = 50) or intervention (n = 50) group. The intervention will be delivered over a period of six months, and with assessments at baseline, and 6 months (end intervention). Upon completion of the RCT, AYLHIV will be randomly selected to participate in two FGDs (n=10 from control group and n=10 from intervention group). AYLHIV in the intervention group will share how the intervention affected their alcohol/drug use as well as their recommendations on how to tailor/improve the intervention to be more culturally appropriate and effective in reducing ADU among AYLHIV in Uganda, while AYLHIV in the control group will share their experiences with ADU risk reduction sessions and how this influenced their ADU.

<u>Description of the control condition:</u> AYLHIV in the control condition will receive ADU risk reduction sessions tailored for AYLHIV. Working with Dr. Mugisha (Consultant), we plan to adapt, expand and tailor the Program for Appropriate Technology in Health (PATH) Life Planning Skills curriculum (Unit 11 on substance use),<sup>232</sup> to

UGANDA VIRUS RESEARCH INSTITUTE
Research Ethics Committee
VALID UNTIL

O3 NOV 2023

APPROVED
P. O. BOX 49, ENTEBBE (U)

include issues specific to AYLHIV. We will train research assistants, using an adapted facilitator's manual, to deliver the adapted curriculum. As part of the RCT, AYLHIV will complete a questionnaire (at baseline and end of the intervention) on their alcohol/drug use behaviors (self-report and biologically measured) and risk/resilience behaviors.

<u>Description of the intervention group</u>: In addition to the adapted ADU training module that the control group will receive, AYLHIV in the intervention arm will receive four (4) Financial Literacy (FL) training sessions and a Youth Development Savings account (YDA) for long-term savings. Although akin to conditional cash transfer interventions, which have become increasingly popular in the social development field by enabling individuals to meet basic needs while incentivizing pro-social behaviors, 132,169,233-235 EE interventions that apply matched savings accounts go beyond incentivizing behavior. They emphasize long-term investment and promote life-long financial inclusion by forming savings habits and establishing partnerships between the participants and local financial institutions and the actual intervention program. For the proposed study, the FEE intervention will be in the form of a YDA, where savings are housed at a local bank and deposits made by the adolescent are matched by the intervention to encourage savings. YDAs yield positive effects, including creating a greater sense of security, self-confidence, and future orientation for young people. 132,169,233-235 Each AYLHIV in the FEE intervention will receive a YDA held in their own name in a bank registered by the Central Bank (Bank of Uganda). We will form partnerships with national banks operating in the study area. . The account will then be matched with money from the program. The maximum Adolescent's contribution to be matched by the program will be an equivalent of US \$20 per month per Adolescent or US \$120 for the 6-month intervention period. Our prior studies indicate that the partner financial institutions have multiple and easily accessible deposit locations in the study area, and that participants can save these amounts. 132,169,233-235 Youth who save the maximum amount will have a total of \$240 at the end of the intervention (\$120 in savings plus \$120 from the match: a 1:1 match). As in the studies that inform this application, each month, a bank account statement will be generated for every AYLHIV to note their accumulated savings. The statements are intended to act as "morale boosters" for the enrolled AYLHIV/ Unique to this study is our innovative spending model, which empowers participants to make informed financial decisions. During the intervention period, AYLHIV will have direct access to both their personal savings deposited in the accounts as well as the match provided by the study. This is different from our prior studies that required the participants' own savings and the match to be kept in separate accounts and to get approval by the research team to access the match. 132,169,233-235 This added unconditional component provides AYLHIV with a safety net to address short-term medical needs and financial and consumption emergencies if they arise. Participants will be provided with financial literacy sessions and mentorship tailored specifically to the needs of AYLHIV and ADU. We expect AYLHIV to be equipped with the knowledge to make well-informed consumption and expenditure decisions, but also feel supported in case of immediate medical needs. The research team will monitor, but not restrict, how participants spend their match. Additionally, the study team will have access to and review participants' bank statements to ascertain deposit and withdrawal frequency. Participants will be encouraged to utilize financial diaries to record their expenditures.

#### C.7.1 Quantitative Data analysis.

Analysis of cross-sectional survey data: Frequency distributions and summary statistics for the outcome and all predictor variables will be derived. The prevalence of ADU from both biological tests and self-reports, assessed using the Smoking and Substance Involvement Screening Test (NIDA-Modified ASSIST)<sup>220</sup> among AYLHIV, will be calculated by dividing the number who tested positive for ADU by the total number of participants tested, and dividing the number screened to be of moderate or high risk in self-reported data by the total number of participants who completed the survey. To determine which multilevel factors are associated with substance misuse, we will fit logistic regression models comprising the outcome (ADU) and potential risk factors with standard errors adjusted for clustering by clinics.

Analysis of RCT data: Primary hypothesis. We hypothesize that participants in the intervention group will have a lower odds of ADU compared to participants in the control group. To test this hypothesis, we will fit three-level mixed-effects models. Each model will comprise the outcome, and fixed categorical effects for study group (intervention vs control), time (baseline, 6-months), and a group-by-time interaction term. Random intercepts will be fitted at the clinic and person level, with unstructured correlations among subjects' repeated measures. Robust Huber-White standard errors and test statistics will be computed for each model. We will assess the omnibus effects for study group, time, and their interaction. Post-estimation analyses will be conducted to assess time-within group simple effects and group within time simple effects. Secondary hypothesis. We hypothesize that AYLHIV in the intervention group will have better mental health outcomes including lower levels of



depressive symptoms, less hopelessness, improved adherence and achieve better viral suppression and improved economic outcomes than AYLHIV in the control group.

### C.7.2. Qualitative data analysis

Interviews will be transcribed and uploaded to QSR NVivo12.<sup>236</sup> Analytic induction techniques<sup>237</sup> will be used for coding. Ten interview transcripts will be randomly selected, read multiple times and independently coded by the team using sensitizing concepts to identify emergent themes (open coding).<sup>238</sup> Broader themes will be broken down into smaller, more specific units until no further subcategory is necessary. Analytic memos will be written to further develop categories, themes, and subthemes, and to integrate the ideas that emerge from the data.<sup>238,239</sup> Codes and the inclusion/exclusion criteria for assigning codes will be discussed as a team to create the final codebook in NVivo. Each transcript will then be independently coded by two investigators using the codebook. Inter-coder reliability will be established. A level of agreement ranging from 66 to 97% based on level of coding indicates good reliability.<sup>240</sup> Disagreements will be resolved through team discussions. The secondary analysis will compare/contrast themes and categories within and across groups to identify similarities, differences, and relationships among findings. Member checking, peer debriefing, and audit trail will be used to ensure rigor.<sup>241</sup>

# C.7.3. Data integration.

The qualitative and quantitative data analyses will be done separately. Findings will be integrated at the interpretation and discussion stages.<sup>242</sup> Conclusions and inferences will be synthesized for a more contextualized and thorough understanding of the multi-level factors associated with ADU among AYLHIV. The mixed methods design will serve two purposes: 1) Complementarity<sup>243,244</sup> and 2) Expansion.<sup>243,244</sup> Qualitative findings will be connected to quantitative findings where the former will provide explanations and context for findings produced by the latter. More specifically, the qualitative data will potentially provide further explanation and contextualization of the local factors that contribute to alcohol and drug abuse among AYLHIV in Uganda. The post-intervention FGDs with AYLHIV who participate in the RCT will explore participants' experiences with the intervention and share recommendations on how it can improve.

# C.8. Potential challenges and alternative strategies.

We do not anticipate major threats to study implementation but we recognize potential concerns. We plan to utilize recruitment strategies that have been successful in ICHAD's NIH funded studies. Should recruitment or enrollment deviate from anticipated rates, we will schedule conference calls to enact solutions and adjust the analytic strategy if necessary.

### C.9. Dissemination.

The research team will facilitate learning across stakeholders and maximize use of the evidence generated through dissemination meetings. Uganda's mental health policy recognizes the burden and impact of ADU on adolescents, their families and communities.<sup>245</sup> If findings warrant, we will leverage these policy guidelines to maximize dissemination of study findings.

#### D. TIMELINE.

First 4 months (April - July 2022) will be spent acquiring IRB, developing/pilot testing study guides and questionnaires, hiring and training project staff, recruiting clinics and selecting participants for the FGDs and QIs. In the next three months (August – October 2022), we will conduct the FGDs and QIs, analyze the transcripts, develop the survey questionnaire concurrently, and then conduct the survey from October and December 2022. Analysis of the quantitative survey will occur from December 2022 to January 2023. Concurrently (from January), we will work on refining the intervention manuals and start recruitment for the 100 participants of the intervention in February 2023. We will allow 8 months to implement the intervention (April– November 2023), giving enough time for follow-up 6 months later. We will conduct the post-intervention FGDs with AYLHIV in December 2023. The rest of the study period will be dedicated to data analysis, preparation of manuscripts, report writing and dissemination.





#### E. REFERENCES

- UNICEF. Adolescent HIV Prevention: HIV in adolescents. 2020;
   https://data.unicef.org/topic/hivaids/adolescents-young-people/. Accessed 06 22 2021, 2021.
- 2. Choudhry V, Agardh A, Stafström M, Östergren P-O. Patterns of alcohol consumption and risky sexual behavior: a cross-sectional study among Ugandan university students. *BMC Public Health*. 2014;14(1):128.
- 3. Walter AW, Lundgren L, Umez-Eronini A, Ritter GA. Alcohol Use and HIV Testing in a National Sample of Women. *AIDS and behavior*. 2016;20 Suppl 1(0 1):S84-S96.
- 4. Bengtson AM, L'Engle K, Mwarogo P, King'ola N. Levels of alcohol use and history of HIV testing among female sex workers in Mombasa, Kenya. *AIDS Care*. 2014;26(12):1619-1624.
- 5. Fatch R, Bellows B, Bagenda F, Mulogo E, Weiser S, Hahn JA. Alcohol Consumption as a Barrier to Prior HIV Testing in a Population-Based Study in Rural Uganda. *AIDS and Behavior*. 2013;17(5):1713-1723.
- 6. Enane LA, Davies M-A, Leroy V, et al. Traversing the cascade: urgent research priorities for implementing the 'treat all' strategy for children and adolescents living with HIV in sub-Saharan Africa. *J Virus Erad.* 2018;4(Suppl 2):40-46.
- 7. Denison JA, Packer C, Stalter RM, et al. Factors Related to Incomplete Adherence to Antiretroviral Therapy among Adolescents Attending Three HIV Clinics in the Copperbelt, Zambia. *AIDS and Behavior*. 2018;22(3):996-1005.
- 8. Kim MH, Mazenga AC, Yu X, et al. High self-reported non-adherence to antiretroviral therapy amongst adolescents living with HIV in Malawi: barriers and associated factors. *Journal of the International AIDS Society.* 2017;20(1):21437.
- 9. Kalichman S, Mathews C, Banas E, Kalichman M. Alcohol-related intentional nonadherence to antiretroviral therapy among people living with HIV, Cape Town, South Africa. *AIDS Care*. 2019;31(8):951-957.
- 10. Haas AD, Technau KG, Pahad S, et al. Mental health, substance use and viral suppression in adolescents receiving ART at a paediatric HIV clinic in South Africa. *J Int AIDS Soc.* 2020;23(12):e25644.
- 11. Petoumenos K, Law MG. Smoking, alcohol and illicit drug use effects on survival in HIV-positive persons. *Curr Opin HIV AIDS*. 2016;11(5):514-520.
- 12. Probst C, Parry CDH, Rehm J. HIV/AIDS mortality attributable to alcohol use in South Africa: a comparative risk assessment by socioeconomic status. *BMJ Open.* 2018;8(2):e017955.
- 13. Cohn SE, Jiang H, McCutchan JA, et al. Association of ongoing drug and alcohol use with non-adherence to antiretroviral therapy and higher risk of AIDS and death: results from ACTG 362. *AIDS Care*. 2011;23(6):775-785.
- 14. UPHIA. UGANDA POPULATION-BASED HIV IMPACT ASSESSMENT UPHIA 2016 | 2017. Uganda2018.
- 15. World Health Organization, Global Health Observatory Data. Total alcohol consumption per capita (liters of pure alcohol, projected estimates, 15+ years of age). In.



- 16. Kuteesa MO, Weiss HA, Cook S, et al. Epidemiology of Alcohol Misuse and Illicit Drug Use Among Young People Aged 15-24 Years in Fishing Communities in Uganda. *Int J Environ Res Public Health*. 2020;17(7):2401.
- 17. Hahn JA, Fatch R, Kabami J, et al. Self-Report of Alcohol Use Increases When Specimens for Alcohol Biomarkers Are Collected in Persons With HIV in Uganda. *JAIDS Journal of Acquired Immune Deficiency Syndromes*. 2012;61(4):e63-e64.
- 18. Hahn JA, Emenyonu NI, Fatch R, et al. Declining and rebounding unhealthy alcohol consumption during the first year of HIV care in rural Uganda, using phosphatidylethanol to augment self-report. *Addiction*. 2016;111(2):272-279.
- 19. Wandera B, Tumwesigye NM, Nankabirwa JI, et al. Alcohol Consumption among HIV-Infected Persons in a Large Urban HIV Clinic in Kampala Uganda: A Constellation of Harmful Behaviors. *PLoS One*. 2015;10(5):e0126236.
- 20. MInistry of Health Uganda. Uganda Population-based HIV Impact Assessment (UPHIA) 2016-2017: Final Report. 2019.
- 21. Kapesa A, Basinda N, Nyanza EC, Mushi MF, Jahanpour O, Ngallaba SE. Prevalence of HIV infection and uptake of HIV/AIDS services among fisherfolk in landing Islands of Lake Victoria, north western Tanzania. BMC Health Serv Res. 2018;18(1):980.
- 22. Smolak A. A meta-analysis and systematic review of HIV risk behavior among fishermen. *AIDS Care.* 2014;26(3):282-291.
- 23. Kissling E, Allison EH, Seeley JA, et al. Fisherfolk are among groups most at risk of HIV: cross-country analysis of prevalence and numbers infected. *AIDS*. 2005;19(17):1939-1946.
- 24. Burke KC, Burke JD, Rae DS, Regier DA. Comparing age at onset of major depression and other psychiatric disorders by birth cohorts in five US community populations. *Archives of general psychiatry*. 1991;48(9):789-795.
- 25. Kessler RC, Angermeyer M, Anthony JC, et al. Lifetime prevalence and age-of-onset distributions of mental disorders in the World Health Organization's World Mental Health Survey Initiative. *World Psychiatry*. 2007;6(3):168-176.
- 26. Kelly TM, Daley DC. Integrated treatment of substance use and psychiatric disorders. *Social work in public health.* 2013;28(3-4):388-406.
- 27. Collins DL, Leibbrandt M. The financial impact of HIV/AIDS on poor households in South Africa. *AIDS* (London, England). 2007.
- 28. Hosegood V, Preston-Whyte E, Busza J, Moitse S, Timaeus IM. Revealing the full extent of households ≥ experiences of HIV and AIDS in rural South Africa. *Social Science & Medicine*. 2007;65(6):1249-1259.
- 29. Masanjala W. The poverty-HIV/AIDS nexus in Africa: a livelihood approach. Social Science & Medicine.

  2007;64(5):1032-1041.

  UGANDA VIRUS RESEARCH INSTITUTE

  VALID UNTIL



- 30. Clark DB, Thatcher DL, Maisto SA. Supervisory neglect and adolescent alcohol use disorders: Effects on AUD onset and treatment outcome. *Addictive Behaviors*. 2005;30(9):1737-1750.
- 31. Eisenberg ME, Toumbourou JW, Catalano RF, Hemphill SA. Social norms in the development of adolescent substance use: a longitudinal analysis of the International Youth Development Study. *J Youth Adolesc.* 2014;43(9):1486-1497.
- 32. El Kazdouh H, El-Ammari A, Bouftini S, El Fakir S, El Achhab Y. Adolescents, parents and teachers 

  perceptions of risk and protective factors of substance use in Moroccan adolescents: a qualitative study.

  Substance Abuse Treatment, Prevention, and Policy. 2018;13(1):31.
- 33. Adeboye A, Yongsong Q, James N. Risky Sexual Behavior and Knowledge of HIV/AIDS among High School Students in Eastern Cape South Africa. *Journal of Human Ecology*. 2016;53(3):194-204.
- 34. Mpofu E, Bility K, Flisher A, Onya H, Lombard C. Correlates of Drug Use in Rural Africa: Drug/Substance Use and Sexual Behaviour in Mankweng District, South Africa. *Journal of Psychology in Africa*. 2005;15:11-15.
- 35. Spear LP. The adolescent brain and age-related behavioral manifestations. *Neuroscience & Biobehavioral Reviews.* 2000;24(4):417-463.
- 36. Mutumba M, Bauermeister JA, Musiime V, et al. Psychosocial challenges and strategies for coping with HIV among adolescents in Uganda: a qualitative study. *AIDS patient care and STDs.* 2015;29(2):86-94.
- 37. Murphy DA, Moscicki AB, Vermund SH, Muenz LR. Psychological distress among HIV+ adolescents in the REACH study: effects of life stress, social support, and coping. *Journal of Adolescent Health*. 2000;27(6):391-398.
- 38. Uebelacker LA, Weisberg RB, Herman DS, Bailey GL, Pinkston-Camp MM, Stein MD. Chronic Pain in HIV-Infected Patients: Relationship to Depression, Substance Use, and Mental Health and Pain Treatment.

  Pain Medicine. 2015;16(10):1870-1881.
- 39. Musisi S, Kinyanda E. Emotional and behavioural disorders in HIV seropositive adolescents in urban Uganda. *East Afr Med J.* 2009;86(1):16-24.
- 40. Adeyemo S, Adeosun II, Ogun OC, et al. Depression and suicidality among adolescents living with human immunodeficiency virus in Lagos, Nigeria. *Child and Adolescent Psychiatry and Mental Health*. 2020;14(1):31.
- 41. Ayano G, Demelash S, Abraha M, Tsegay L. The prevalence of depression among adolescent with HIV/AIDS: a systematic review and meta-analysis. *AIDS Research and Therapy.* 2021;18(1):23.
- 42. Cavazos-Rehg P, Xu C, Borodovsky J, et al. The impact of discomfort with HIV status and hopelessness on depressive symptoms among adolescents living with HIV in Uganda. *AIDS Care*. 2021;33(7):867-872.
- 43. Cooper ML, Kuntsche E, Levitt A, Barber LL, Wolf S. Motivational models of substance use: A review of theory and research on motives for using alcohol, marijuana, and tobacco. In: *The Oxford handbook of substance use and substance use disorders, Vol. 1.* New York, NY, US: Oxford University Press; 2016:375-421.

  UGANDA VIRUS RESEARCH INSTITUTE
  Research Ethics Committee
  VALID UNTIL

- 44. Cooper ML. Motivations for alcohol use among adolescents: Development and validation of a four-factor model. *Psychological Assessment*. 1994;6(2):117-128.
- 45. Cooper ML, Frone MR, Russell M, Mudar P. Drinking to regulate positive and negative emotions: A motivational model of alcohol use. *Journal of Personality and Social Psychology.* 1995;69(5):990-1005.
- 46. Sayette MA. Does drinking reduce stress? *Alcohol Research & Health.* 1999;23(4):250-250.
- 47. Bandura A. A sociocognitive analysis of substance abuse: An agentic perspective. *Psychological science*. 1999;10(3):214-217.
- 48. Kuria MW, Ndetei DM, Obot IS, et al. The Association between Alcohol Dependence and Depression before and after Treatment for Alcohol Dependence. *ISRN Psychiatry*. 2012;2012:482802-482802.
- 49. McHugh RK, Weiss RD. Alcohol Use Disorder and Depressive Disorders. *Alcohol Res.* 2019;40(1):arcr.v40.41.01.
- 50. Nabyonga-Orem J, Bazeyo W, Okema A, Karamagi H, Walker O. Effect of HIV/AIDS on household welfare in Uganda rural communities: a review. *East Afr Med J.* 2008;85(4):187-196.
- 51. Cerdá M, Diez-Roux AV, Tchetgen ET, Gordon-Larsen P, Kiefe C. The relationship between neighborhood poverty and alcohol use: estimation by marginal structural models. *Epidemiology*. 2010;21(4):482-489.
- 52. Gavin L, Galavotti C, Dube H, et al. Factors associated with HIV infection in adolescent females in Zimbabwe. *Journal of Adolescent Health.* 2006;39(4):596. e511-596. e518.
- 53. Jaspan HB, Berwick JR, Myer L, et al. Adolescent HIV prevalence, sexual risk, and willingness to participate in HIV vaccine trials. *Journal of adolescent health.* 2006;39(5):642-648.
- Test F, Mehta S, Handler A, Mutimura E, Bamukunde A, Cohen M. Gender inequities in sexual risks among youth with HIV in Kigali, Rwanda. *International journal of STD & AIDS*. 2012;23(6):394-399.
- 55. Ssewanyana D, Mwangala PN, Van Baar A, Newton CR, Abubakar A. Health risk behaviour among adolescents living with HIV in sub-Saharan Africa: a systematic review and meta-analysis. *BioMed research international*. 2018;2018.
- 56. Hawkins JD, Arthur MW, Catalano RF. Preventing substance abuse. *Crime and justice*. 1995;19:343-427.
- 57. Ogundipe O, Amoo E, Adeloye D, Olawole-Isaac A. Substance use among adolescents in sub-Saharan Africa: A systematic review and meta-analysis. *South African Journal of Child Health.* 2018;2018(1):s79-s84.
- 58. World Health Organization. *Global status report on alcohol and health 2018.* World Health Organization; 2019.
- 59. Culbreth R, Masyn KE, Swahn MH, Self-Brown S, Kasirye R. The interrelationships of child maltreatment, alcohol use, and suicidal ideation among youth living in the slums of Kampala, Uganda. *Child Abuse Negl.* 2021;112:104904.





- 60. Kabwama SN, Matovu JKB, Ssenkusu JM, Ssekamatte T, Wanyenze RK. Alcohol use and associated factors among adolescent boys and young men in Kampala, Uganda. *Substance Abuse Treatment, Prevention, and Policy.* 2021;16(1):49.
- 61. Kiene SM, Sileo KM, Dove M, Kintu M. Hazardous alcohol consumption and alcohol-related problems are associated with unknown and HIV-positive status in fishing communities in Uganda. *AIDS Care*. 2019;31(4):451-459.
- 62. Tumwesigye NM, Atuyambe L, Wanyenze RK, et al. Alcohol consumption and risky sexual behaviour in the fishing communities: evidence from two fish landing sites on Lake Victoria in Uganda. *BMC public health*. 2012;12(1):1-11.
- 63. Breuer C, Bloom B, Miller AP, et al. <sub>Φ</sub>The Bottle Is My Wife <sub>Φ</sub>: Exploring Reasons Why Men Drink Alcoho in Ugandan Fishing Communities. *Social Work in Public Health*. 2019;34(8):657-672.
- 64. Wandera SO, Tumwesigye NM, Walakira EJ, Kisaakye P, Wagman J. Alcohol use, intimate partner violence, and HIV sexual risk behavior among young people in fishing communities of Lake Victoria, Uganda. *BMC Public Health*. 2021;21(1):544.
- 65. Jewkes R, Dunkle K, Nduna M, et al. Factors associated with HIV sero-status in young rural South African women: connections between intimate partner violence and HIV. *International journal of epidemiology*. 2006;35(6):1461-1468.
- 66. Jewkes R, Dunkle K, Nduna M, et al. Factors associated with HIV sero-positivity in young, rural South African men. *International journal of epidemiology*. 2006;35(6):1455-1460.
- 67. Birungi C, Ssembajjwe W, Salisbury T, et al. Substance use among HIV-infected adolescents in Uganda: rates and association with potential risks and outcome factors. *AIDS care*. 2021;33(2):137-147.
- 68. Kresina TF, Lubran R. The Linkage of Illicit Drug Use / Alcohol Use and HIV Infection in Young Adults. *Int J High Risk Behav Addict*. 2017;6(1):e32129.
- 69. Doku D. Substance use and risky sexual behaviours among sexually experienced Ghanaian youth. *BMC Public Health.* 2012;12(1):571.
- 70. Pufall EL, Eaton JW, Robertson L, Mushati P, Nyamukapa C, Gregson S. Education, substance use, and HIV risk among orphaned adolescents in Eastern Zimbabwe. *Vulnerable Children and Youth Studies*. 2017;12(4):360-374.
- 71. Seff I, Steiner JJ, Stark L. Early sexual debut: A multi-country, sex-stratified analysis in sub-Saharan Africa. *Global Public Health*. 2021;16(7):1046-1056.
- 72. Woolf-King SE, Maisto SA. Alcohol use and high-risk sexual behavior in Sub-Saharan Africa: a narrative review. *Arch Sex Behav.* 2011;40(1):17-42.
- 73. Baliunas D, Rehm J, Irving H, Shuper P. Alcohol consumption and risk of incident human immunodeficiency virus infection: a meta-analysis. *Int J Public Health.* 2010;55(3):159-166.





- 74. Barhafumwa B, Dietrich J, Closson K, et al. High prevalence of depression symptomology among adolescents in Soweto, South Africa associated with being female and cofactors relating to HIV transmission. *Vulnerable Children and Youth Studies*. 2016;11(3):263-273.
- 75. Magidson JF, Dietrich J, Otwombe KN, Sikkema KJ, Katz IT, Gray GE. Psychosocial correlates of alcohol and other substance use among low-income adolescents in peri-urban Johannesburg, South Africa: A focus on gender differences. *Journal of Health Psychology*. 2017;22(11):1415-1425.
- 76. Nalugya-Sserunjogi J, Rukundo GZ, Ovuga E, Kiwuwa SM, Musisi S, Nakimuli-Mpungu E. Prevalence and factors associated with depression symptoms among school-going adolescents in Central Uganda. *Child Adolesc Psychiatry Ment Health.* 2016;10(1):39.
- 77. Oppong Asante K, Kugbey N. Alcohol use by school-going adolescents in Ghana: Prevalence and correlates. *Mental Health and Prevention*. 2019;13:75-81.
- 78. Kessler RC, Amminger GP, Aguilar-Gaxiola S, Alonso J, Lee S, Ustun TB. Age of onset of mental disorders: a review of recent literature. *Current opinion in psychiatry*. 2007;20(4):359.
- 79. Cupp PK, Zimmerman RS, Bhana A, et al. Combining and adapting American school-based alcohol and HIV prevention programmes in South Africa: The HAPS project. *Vulnerable Children and Youth Studies*. 2008;3(2):134-142.
- 80. Francis JM, Myers B, Nkosi S, et al. The prevalence of religiosity and association between religiosity and alcohol use, other drug use, and risky sexual behaviours among grade 8-10 learners in Western Cape, South Africa. *PloS one*. 2019;14(2):e0211322.
- 81. McGill E, Petticrew M, Marks D, McGrath M, Rinaldi C, Egan M. Applying a complex systems perspective to alcohol consumption and the prevention of alcohol-related harms in the 21st century: a scoping review. *Addiction*. 2021.
- 82. Nyundo A, Manu A, Regan M, et al. Factors associated with depressive symptoms and suicidal ideation and behaviours amongst sub-Saharan African adolescents aged 10-19 years: cross-sectional study.

  \*Tropical Medicine & International Health. 2020;25(1):54-69.
- 83. Schulenberg JE, Maggs JL. A developmental perspective on alcohol use and heavy drinking during adolescence and the transition to young adulthood. *Journal of Studies on Alcohol, Supplement*. 2002(14):54-70.
- 84. Wallace Jr JM, Yamaguchi R, Bachman JG, O'Malley PM, Schulenberg JE, Johnston LD. Religiosity and adolescent substance use: The role of individual and contextual influences. *Social problems*. 2007;54(2):308-327.
- 85. Brooks-Russell A, Simons-Morton B, Haynie D, Farhat T, Wang J. Longitudinal relationship between drinking with peers, descriptive norms, and adolescent alcohol use. *Prevention science*. 2014;15(4):497-505.
- 86. Bouchard M, Gallupe O, Dawson K, Anamali M. No place like home? Availability, opportunity, and substance use in adolescence. *Journal of Youth Studies*. 2018;21(6):747-764.



15

- 87. Ghuman S, Meyer-Weitz A, Knight S. Prevalence patterns and predictors of alcohol use and abuse among secondary school students in southern KwaZulu-Natal, South Africa: demographic factors and the influence of parents and peers. *South African Family Practice*. 2012;54(2):132-138.
- 88. Leung RK, Toumbourou JW, Hemphill SA. The effect of peer influence and selection processes on adolescent alcohol use: a systematic review of longitudinal studies. *Health psychology review*. 2014;8(4):426-457.
- 89. Manu E, Douglas M, Ntsaba MJ. Contextual influences of illicit adolescent marijuana cultivation and trading in the Inqguza Hill local municipality of South Africa: implications for public health policy. *Substance abuse treatment, prevention, and policy.* 2021;16(1):1-15.
- 90. Muchiri BW, Dos Santos MM. Family management risk and protective factors for adolescent substance use in South Africa. *Substance abuse treatment, prevention, and policy.* 2018;13(1):1-10.
- 91. Obadeji A, Kumolalo BF, Oluwole LO, Ajiboye AS, Dada MU, Ebeyi RC. Substance use among adolescent high school students in Nigeria and its relationship with psychosocial factors. *Journal of Research in Health Sciences*. 2020;20(2):e00480.
- 92. Ogunsola OO, Fatusi AO. Risk and protective factors for adolescent substance use: a comparative study of secondary school students in rural and urban areas of Osun State, Nigeria. *International Journal of Adolescent Medicine and Health.* 2017;29(3).
- 93. Ryan SM, Jorm AF, Lubman DI. Parenting factors associated with reduced adolescent alcohol use: a systematic review of longitudinal studies. *Australian & New Zealand Journal of Psychiatry*. 2010;44(9):774-783.
- 94. Tyler KA, Handema R, Schmitz RM, Phiri F, Kuyper KS, Wood C. Multi-level risk and protective factors for substance use among Zambian street youth. *Substance use & misuse*. 2016;51(7):922-931.
- 95. Yap MB, Cheong TW, Zaravinos-Tsakos F, Lubman DI, Jorm AF. Modifiable parenting factors associated with adolescent alcohol misuse: a systematic review and meta-analysis of longitudinal studies. *Addiction*. 2017;112(7):1142-1162.
- 96. Kang E, Mellins CA, Dolezal C, Elkington KS, Abrams EJ. Disadvantaged neighborhood influences on depression and anxiety in youth with perinatally acquired human immunodeficiency virus: how life stressors matter. *Journal of community psychology*. 2011;39(8):956-971.
- 97. Mellins CA, Malee KM. Understanding the mental health of youth living with perinatal HIV infection: lessons learned and current challenges. *J Int AIDS Soc.* 2013;16:18593.
- 98. Mutumba M, Bauermeister JA, Musiime V, et al. Psychosocial challenges and strategies for coping with HIV among adolescents in Uganda: a qualitative study. *AIDS patient care and STDs.* 2014.
- 99. Scharko A. DSM psychiatric disorders in the context of pediatric HIV/AIDS. *AIDS care*. 2006;18(5):441-445.
- 100. Brown LK, Whiteley L, Harper GW, Nichols S, Nieves A. Psychological Symptoms Among 2032 Youth Living with HIV: A Multisite Study. *AIDS patient care and STDs.* 2015.





- 101. Malee KM, Tassiopoulos K, Huo Y, et al. Mental health functioning among children and adolescents with perinatal HIV infection and perinatal HIV exposure. *AIDS Care*. 2011;23(12):1533-1544.
- 102. Louthrenoo O, Oberdorfer P, Sirisanthana V. Psychosocial functioning in adolescents with perinatal HIV infection receiving highly active antiretroviral therapy. *Journal of the International Association of Providers of AIDS Care (JIAPAC)*. 2013:2325957413488171.
- 103. Kessler RC, Aguilar-Gaxiola S, Andrade L, et al. Mental-substance comorbidities in the ICPE surveys. 2014.
- 104. Elkington KS, Bauermeister JA, Zimmerman MA. Psychological distress, substance use, and HIV/STI risk behaviors among youth. *J Youth Adolesc.* 2010;39(5):514-527.
- 105. Williams PL, Leister E, Chernoff M, et al. Substance use and its association with psychiatric symptoms in perinatally HIV-infected and HIV-affected adolescents. *AIDS Behav.* 2010;14(5):1072-1082.
- 106. Dessauvagie AS, Jörns-Presentati A, Napp AK, et al. The prevalence of mental health problems in sub-Saharan adolescents living with HIV: a systematic review. *Global Mental Health*. 2020;7:e29.
- 107. Malee KM, Tassiopoulos K, Huo Y, et al. Mental health functioning among children and adolescents with perinatal HIV infection and perinatal HIV exposure. *AIDS care*. 2011;23(12):1533-1544.
- 108. Remien RH, Stirratt MJ, Nguyen N, Robbins RN, Pala AN, Mellins CA. Mental health and HIV/AIDS: the need for an integrated response. *AIDS (London, England)*. 2019;33(9):1411.
- 109. Vreeman RC, McCoy BM, Lee S. Mental health challenges among adolescents living with HIV. *Journal of the International AIDS Society.* 2017;20:21497.
- 110. Woollett N, Cluver L, Bandeira M, Brahmbhatt H. Identifying risks for mental health problems in HIV positive adolescents accessing HIV treatment in Johannesburg. *Journal of Child & Adolescent Mental Health*. 2017;29(1):11-26.
- 111. Mellins CA, Brackis-Cott E, Dolezal C, Abrams EJ. The role of psychosocial and family factors in adherence to antiretroviral treatment in human immunodeficiency virus-infected children. *The Pediatric infectious disease journal*. 2004;23(11):1035-1041.
- 112. Mellins CA, Tassiopoulos K, Malee K, et al. Behavioral health risks in perinatally HIV-exposed youth: co-occurrence of sexual and drug use behavior, mental health problems, and nonadherence to antiretroviral treatment. *AIDS Patient Care STDS*. 2011;25(7):413-422.
- 113. Naar-King S, Templin T, Wright K, Frey M, Parsons JT, Lam P. Psychosocial factors and medication adherence in HIV-positive youth. *AIDS Patient Care & STDs.* 2006;20(1):44-47.
- 114. Elkington KS, Bauermeister JA, Santamaria EK, Dolezal C, Mellins CA. Substance Use and the Development of Sexual Risk Behaviors in Youth Perinatally Exposed to HIV. *Journal of pediatric psychology*. 2014.
- 115. Elkington KS, Teplin LA, Mericle AA, Welty LJ, Romero EG, Abram KM. HIV/sexually transmitted infection risk behaviors in delinquent youth with psychiatric disorders: a longitudinal study. *Journal of the American Academy of Child and Adolescent Psychiatry*. 2008;47(8):901-911.



- 116. Fair C, Wiener L, Zadeh S, et al. Reproductive health decision-making in perinatally HIV-infected adolescents and young adults. *Maternal and child health journal*. 2013;17(5):797-808.
- 117. Wilson DP, Law MG, Grulich AE, Cooper DA, Kaldor JM. Relation between HIV viral load and infectiousness: a model-based analysis. *The Lancet*. 2008;372(9635):314-320.
- 118. Bangsberg DR. Preventing HIV antiretroviral resistance through better monitoring of treatment adherence. *Journal of Infectious Diseases*. 2008;197(Supplement 3):S272-S278.
- 119. Little SJ, Holte S, Routy J-P, et al. Antiretroviral-drug resistance among patients recently infected with HIV. *New England Journal of Medicine*. 2002;347(6):385-394.
- 120. Jörns-Presentati A, Napp A-K, Dessauvagie AS, et al. The prevalence of mental health problems in sub-Saharan adolescents: A systematic review. *PLOS ONE*. 2021;16(5):e0251689.
- 121. Marwick KF, Kaaya SF. Prevalence of depression and anxiety disorders in HIV-positive outpatients in rural Tanzania. *AIDS Care*. 2010;22(4):415-419.
- 122. Marais BJ, Esser M, Godwin S, Rabie H, Cotton MF. Poverty and human immunodeficiency virus in children: a view from the Western Cape, South Africa. *Annals of the New York Academy of Sciences*. 2008;1136(1):21-27.
- 123. Bermudez LG, Ssewamala FM, Neilands TB, et al. Does economic strengthening improve viral suppression among adolescents living with HIV? Results from a cluster randomized trial in Uganda. *J AIDS & Behavior.* 2018;22(11):3763-3772.
- 124. Ssewamala FM, Dvalishvili D, Mellins CA, et al. The long-term effects of a family based economic empowerment intervention (Suubi+ Adherence) on suppression of HIV viral loads among adolescents living with HIV in southern Uganda: Findings from 5-year cluster randomized trial. *PLOS ONE*. 2020;15(2):e0228370.
- 125. Ramadhani HO, Thielman NM, Landman KZ, et al. Predictors of incomplete adherence, virologic failure, and antiviral drug resistance among HIV-infected adults receiving antiretroviral therapy in Tanzania. *Clinical Infectious Diseases*. 2007;45(11):1492-1498.
- Tuller DM, Bangsberg DR, Senkungu J, Ware NC, Emenyonu N, Weiser SD. Transportation costs impede sustained adherence and access to HAART in a clinic population in southwestern Uganda: a qualitative study. *AIDS & Behavior*. 2010;14(4):778-784.
- 127. Weiser S, Wolfe W, Bangsberg D, et al. Barriers to antiretroviral adherence for patients living with HIV infection and AIDS in Botswana. *AIDS (London, England)*. 2003;34(3):281-288.
- Weiser SD, Tuller DM, Frongillo EA, Senkungu J, Mukiibi N, Bangsberg DR. Food insecurity as a barrier to sustained antiretroviral therapy adherence in Uganda. *PLOS ONE*. 2010;5(4):e10340.
- 129. Young S, Wheeler AC, McCoy SI, Weiser SD. A review of the role of food insecurity in adherence to care and treatment among adult and pediatric populations living with HIV and AIDS. *AIDS & Behavior*. 2014;18(5):505-515.



- 130. Lund C, Breen A, Flisher AJ, et al. Poverty and common mental disorders in low and middle income countries: A systematic review. *Social Science & Medicine*. 2010;71(3):517-528.
- 131. Nabunya P, Ssewamala FM, Ilic V. Family economic strengthening and parenting stress among caregivers of AIDS-orphaned children: results from a cluster randomized clinical trial in Uganda. *Children and Youth Services Review.* 2014;44:417-421.
- 132. Ismayilova L, Ssewamala FM, Karimli L. Family support as a mediator of change in sexual risk-taking attitudes among orphaned adolescents in rural Uganda. *Journal of Adolescent Health.* 2012;50(3):228-235.
- 133. Ssewamala FM, Karimli L, Han C-K, Ismayilova L. Social capital, savings, and educational performance of orphaned adolescents in Sub-Saharan Africa. *Children and Youth Services Review.* 2010;32(12):1704-1710.
- 134. Ismayilova L, Karimli L. Harsh parenting and violence against children: a trial with ultrapoor families in Francophone West Africa. *Journal of Clinical Child & Adolescent Psychology.* 2020;49(1):18-35.
- 135. Lachman J, Spreckelsen TF, Wamoyi J, Wight D, Maganga J, Gardner F. Combining Economic Strengthening and Parenting Programmes to Reduce Violence Against Children in Rural Tanzania: A Cluster Randomised Controlled Trial. *BMJ Global Health*. 2020.
- 136. Amerikaner M, Monks G, Wolfe P, Thomas S. Family interaction and individual psychological health. *%J Journal of Counseling Development*. 1994;72(6):614-620.
- 137. Kotchick BA, Dorsey S, Miller KS, Forehand R. Adolescent sexual risk-taking behavior in single-parent ethnic minority families. *Journal of Family Psychology*. 1999;13(1):93.
- 138. McNeely C, Shew ML, Beuhring T, Sieving R, Miller BC, Blum RW. Mothers ← influence on the timing of first sex among 14-and 15-year-olds. *Journal of Adolescent Health*. 2002;31(3):256-265.
- 139. Miller KS, Forehand R, Kotchick BA. Adolescent sexual behavior in two ethnic minority samples: The role of family variables. *Journal of Marriage and the Family*. 1999:85-98.
- 140. Resnick MD, Bearman PS, Blum RW, et al. Protecting adolescents from harm: findings from the National Longitudinal Study on Adolescent Health. *JAMA*. 1997;278(10):823-832.
- 141. Jewkes R, Nduna M, Levin J, et al. Impact of stepping stones on incidence of HIV and HSV-2 and sexual behaviour in rural South Africa: cluster randomised controlled trial. *Bmj.* 2008;337.
- 142. Carney T, Browne FA, Myers B, Kline TL, Howard B, Wechsberg WM. Adolescent female school dropouts who use drugs and engage in risky sex: Effects of a brief pilot intervention in Cape Town, South Africa.

  AIDS care. 2019;31(1):77-84.
- 143. Carney T, Johnson K, Carrico A, Myers B. Acceptability and feasibility of a brief substance use intervention for adolescents in Cape Town, South Africa: A pilot study. *International journal of psychology.* 2020;55(6):1016-1025.
- 144. Cluver L, Meinck F, Yakubovich A, et al. Reducing child abuse amongst adolescents in low-and middle-income countries: A pre-post trial in South Africa. *BMC public health*. 2016;16(1):1-11.





- 145. Jemmott III JB, Jemmott LS, O∝Leary A, et al. Cognitive-behavioural health-promotion intervention increases fruit and vegetable consumption and physical activity among South African adolescents: a cluster-randomised controlled trial. *Psychology and Health*. 2011;26(2):167-185.
- 146. Motamedi M, Caldwell L, Wegner L, Smith E, Jones D. Girls just want to know where to have fun: Preventing substance use initiation in an under-resourced community in South Africa through HealthWise. *Prevention science*. 2016;17(6):700-709.
- 147. Resnicow K, Reddy SP, James S, et al. Comparison of two school-based smoking prevention programs among South African high school students: results of a randomized trial. *Annals of Behavioral Medicine*. 2008;36(3):231-243.
- 148. Smith EA, Palen L-A, Caldwell LL, et al. Substance use and sexual risk prevention in Cape Town, South Africa: an evaluation of the HealthWise program. *Prevention Science*. 2008;9(4):311-321.
- 149. Tibbits MK, Smith EA, Caldwell LL, Flisher AJ. Impact of HealthWise South Africa on polydrug use and high-risk sexual behavior. *Health education research*. 2011;26(4):653-663.
- 150. Bermudez LG, Jennings L, Ssewamala FM, Nabunya P, Mellins C, McKay M. Equity in adherence to antiretroviral therapy among economically vulnerable adolescents living with HIV in Uganda. *J African journal of AIDS Research.* 2016;28(sup2):83-91.
- 151. Han C-K, Ssewamala FM, Wang JS-H. Family economic empowerment and mental health among AIDS-affected children living in AIDS-impacted communities: evidence from a randomised evaluation in southwestern Uganda. *J Epidemiol Community Health*. 2013;67(3):225-230.
- 152. Jennings L, Ssewamala FM, Nabunya P. Effect of savings-led economic empowerment on HIV preventive practices among orphaned adolescents in rural Uganda: results from the Suubi-Maka randomized experiment. *AIDS care*. 2016;28(3):273-282.
- 153. Ssewamala FM, Han C-K, Neilands TB, Ismayilova L, Sperber E. Effect of economic assets on sexual risk-taking intentions among orphaned adolescents in Uganda. *American Journal of Public Health*. 2010;100(3):483-488.
- 154. Bronfenbrenner U. Ecological models of human development. *Readings on the development of children.* 1994;2(1):37-43.
- 155. Earnshaw VA, Chaudoir SR. From conceptualizing to measuring HIV stigma: a review of HIV stigma mechanism measures. *J AIDS & Behavior*. 2009;13(6):1160.
- 156. Ssewamala FM, Sperber E, Zimmerman JM, Karimli L. The potential of asset-based development strategies for poverty alleviation in Sub-Saharan Africa. *International Journal of Social Welfare*. 2010;19(4):433-443.
- 157. Sherraden M. Assets and the poor: A new American welfare policy. . In. New York: ME Sharpe; 1991.
- 158. Zimmerman GM, Farrell C. Parents, peers, perceived risk of harm, and the neighborhood: Contextualizing key influences on adolescent substance use. *J Youth Adolesc.* 2017;46(1):228-247.





- 159. Elkington KS, Bauermeister JA, Zimmerman MA. Do parents and peers matter? A prospective socioecological examination of substance use and sexual risk among African American youth. *Journal of adolescence*. 2011;34(5):1035-1047.
- 160. Jacobs W, Amuta-Jimenez AO, Olusanya OA, Bristow AF, Adeloye D, Barry AE. Socio-ecological factors of adolescent substance use in Nigeria: a systematic review of literature. *Journal of health care for the poor and underserved.* 2020;31(4):1765-1784.
- 161. Scribner R, Theall KP, Simonsen N, Robinson W. HIV risk and the alcohol environment: advancing an ecological epidemiology for HIV/AIDS. *Alcohol Research & Health*. 2010;33(3):179.
- 162. Ssewanyana D, Mwangala PN, Marsh V, et al. Socio-ecological determinants of alcohol, tobacco, and drug use behavior of adolescents in Kilifi County at the Kenyan coast. *Journal of health psychology*. 2020;25(12):1940-1953.
- 163. Dohrenwend BP, Levav I, Shrout PE, et al. Socioeconomic status and psychiatric disorders: the causation-selection issue. *Science*. 1992;255(5047):946-952.
- 164. Wagman JA, Nabukalu D, Miller AP, et al. Prevalence and correlates of men ∠s and women ∠s alcoho use in agrarian, trading and fishing communities in Rakai, Uganda. *PLOS ONE*. 2020;15(10):e0240796.
- 165. Naamara W, Muhwezi WW. Factors Associated With Alcohol Dependence Among Adult Male Clients in Butabika Hospital, Uganda. *Journal of Social Work Practice in the Addictions*. 2014;14(3):322-326.
- 166. Jones SE, Underwood JM, Pampati S, et al. School-level poverty and persistent feelings of sadness or hopelessness, suicidality, and experiences with violence victimization among public high school students. *Journal of health care for the poor and underserved.* 2020;31(3):1248-1263.
- 167. Reiss F. Socioeconomic inequalities and mental health problems in children and adolescents: A systematic review. *Social Science & Medicine*. 2013;90:24-31.
- 168. Sherraden M. Stakeholding: Notes on a Theory of Welfare Based on Assets. *Social Service Review*. 1990;64(4):580-601.
- 169. Han C-K, Ssewamala FM, Wang JS-H. Family economic empowerment and mental health among AIDS-affected children living in AIDS-impacted communities: evidence from a randomised evaluation in southwestern Uganda. *Journal of Epidemiology and Community Health*. 2013;67(3):225-230.
- 170. Cavazos-Rehg P, Byansi W, Xu C, et al. The Impact of a Family-Based Economic Intervention on the Mental Health of HIV-Infected Adolescents in Uganda: Results From Suubi + Adherence. *J Adolesc Health*. 2021;68(4):742-749.
- 171. Greenfield TK, Kerr WC. Alcohol measurement methodology in epidemiology: recent advances and opportunities. *Addiction*. 2008;103(7):1082-1099.
- 172. Dawson D. Methodological Issues in Measuring Alcohol Use. 2003; https://pubs.niaaa.nih.gov/publications/arh27-1/18-29.htm. Accessed 7/20, 2021.
- 173. Sserunjogi B. Alcohol Consumption among Youth in Uganda: Why Policy Intervention Is Necessary. *YOUTH FOR POLICY PERSPECTIVES.* 2018;6(13.5):14.





- 174. Brathwaite R, Rocha TB-M, Kieling C, et al. Predicting the risk of depression among adolescents in Nepal using a model developed in Brazil: the IDEA Project. *European Child & Adolescent Psychiatry*. 2020.
- 175. Brathwaite R, Rocha TB-M, Kieling C, et al. Predicting the risk of future depression among school-attending adolescents in Nigeria using a model developed in Brazil. *Psychiatry Research*. 2020;294:113511.
- 176. Brathwaite R, Ssewamala FM, Neilands TB, Nabunya P, Byansi W, Damulira C. Development and external validation of a risk calculator to predict internalising symptoms among Ugandan youths affected by HIV. *Psychiatry Research.* 2021;302:114028.
- 177. Harris M, Brathwaite R, McGowan CR, et al. 'Care and Prevent': rationale for investigating skin and soft tissue infections and AA amyloidosis among people who inject drugs in London. *Harm Reduct J.* 2018;15(1):23.
- 178. Harris M, Brathwaite R, Scott J, et al. Drawing attention to a neglected injecting-related harm: a systematic review of AA amyloidosis among people who inject drugs. *Addiction*. 2018;113(10):1790-1801.
- 179. Harris M, Scott J, Wright T, Brathwaite R, Ciccarone D, Hope V. Injecting-related health harms and overuse of acidifiers among people who inject heroin and crack cocaine in London: a mixed-methods study. *Harm Reduction Journal*. 2019;16(1):60.
- 180. McGowan CR, Wright T, Nitsch D, et al. High prevalence of albuminuria amongst people who inject drugs: A cross-sectional study. *Scientific Reports*. 2020;10(1):7059.
- 181. Brathwaite R, Addo J, Kunst AE, et al. Smoking prevalence differs by location of residence among Ghanaians in Africa and Europe: The RODAM study. *PLOS ONE*. 2017;12(5):e0177291.
- 182. Brathwaite R, Addo J, Smeeth L, Lock K. A Systematic Review of Tobacco Smoking Prevalence and Description of Tobacco Control Strategies in Sub-Saharan African Countries; 2007 to 2014. *PLoS One.* 2015;10(7):e0132401.
- 183. Brathwaite R, Smeeth L, Addo J, et al. Ethnic differences in current smoking and former smoking in the Netherlands and the contribution of socioeconomic factors: a cross-sectional analysis of the HELIUS study. *BMJ Open.* 2017;7(7):e016041.
- 184. Maharaj RG, Babwah T, Motilal MS, et al. The National Alcohol Survey of Households in Trinidad and Tobago (NASHTT): willingness to support changes in policy, laws and regulations. *BMC Public Health*. 2018;18(1):1202.
- 185. Maharaj RG, Motilal MS, Babwah T, et al. National Alcohol Survey of households in Trinidad and Tobago (NASHTT): Alcohol use in households. *BMC Public Health*. 2017;17(1):347.
- 186. Ssewamala FM, Shu-Huah Wang J, Brathwaite R, et al. Impact of a Family Economic Intervention (Bridges) on Health Functioning of Adolescents Orphaned by HIV/AIDS: A 5-Year (2012 <sub>1</sub> 2017) Cluster Randomized Controlled Trial in Uganda. *Am J Public Health*. 2021:e1-e10.
- 187. Weiser SD, Palar K, Frongillo EA, et al. Longitudinal assessment of associations between food insecurity, antiretroviral adherence and HIV treatment outcomes in rural Uganda. *AIDS (London, England)*. 2014;28(1):115-120.



- 188. Musiime V, Kasirye P, Naidoo-James B, et al. Once vs twice-daily abacavir and lamivudine in African children. *AIDS (London, England)*. 2016;30(11):1761-1770.
- 189. Kwansah J, Dzodzomenyo M, Mutumba M, et al. Policy talk: incentives for rural service among nurses in Ghana. *Health Policy and Planning*. 2012;27(8):669-676.
- 190. Snow RC, Asabir K, Mutumba M, et al. Key factors leading to reduced recruitment and retention of health professionals in remote areas of Ghana: a qualitative study and proposed policy solutions. *Human resources for health.* 2011;9(1):13.
- 191. Mutumba M, Bauermeister JA, Elkington KS, et al. A prospective longitudinal study of mental health symptoms among perinatally HIV-infected and HIV-exposed but uninfected urban youths. *Journal of Adolescent Health*. 2016;58(4):460-466.
- 192. Mutumba M, Bauermeister JA, Harper GW, et al. Psychological distress among Ugandan adolescents living with HIV: Examining stressors and the buffering role of general and religious coping strategies. *Global public health.* 2017;12(12):1479-1491.
- 193. Mutumba M, Harper GW. Mental health and support among young key populations: an ecological approach to understanding and intervention. *J Int AIDS Soc.* 2015;18:19429.
- 194. Mutumba M, Musiime V, Lepkwoski JM, et al. Examining the relationship between psychological distress and adherence to anti-retroviral therapy among Ugandan adolescents living with HIV. *AIDS care*. 2016;28(7):807-815.
- 195. Mutumba M, Musiime V, Tsai AC, et al. Disclosure of HIV status to perinatally infected adolescents in urban Uganda: a qualitative study on timing, process, and outcomes. *Journal of the Association of Nurses in AIDS Care.* 2015;26(4):472-484.
- 196. Mutumba M, Tomlinson M, Tsai AC. Psychometric properties of instruments for assessing depression among African youth: A systematic review. *Journal of child and adolescent mental health*. 2014;26(2):139-156.
- 197. Filiatreau LM, Ebasone PV, Dzudie A, et al. Correlates of self-reported history of mental health help-seeking: a cross-sectional study among individuals with symptoms of a mental or substance use disorder initiating care for HIV in Cameroon. *BMC Psychiatry*. 2021;21(1):293.
- 198. Filiatreau LM, Giovenco D, Twine R, et al. Examining the relationship between physical and sexual violence and psychosocial health in young people living with HIV in rural South Africa. *Journal of the International AIDS Society.* 2020;23(12):e25654.
- 199. Filiatreau LM, Pettifor A, Edwards JK, et al. Associations Between Key Psychosocial Stressors and Viral Suppression and Retention in Care Among Youth with HIV in Rural South Africa. *AIDS Behav.* 2021;25(8):2358-2368.
- 200. Filiatreau LM, Wright M, Kimaru L, et al. Correlates of ART Use Among Newly Diagnosed HIV Positive Adolescent Girls and Young Women Enrolled in HPTN 068. *AIDS Behav.* 2020;24(9):2606-2615.





- 201. Pettifor A, Filiatreau L, Delany-Moretlwe S. Time to strengthen HIV treatment and prevention for youth. *The Lancet HIV.* 2019;6(11):e727-e728.
- 202. Parcesepe AM, Filiatreau LM, Ebasone PV, et al. Gender, Mental Health, and Entry Into Care with Advanced HIV Among People Living with HIV in Cameroon Under a National 'Treat All' Policy. *AIDS Behav.* 2021.
- 203. Edwards JK, Cole SR, Breger TL, et al. Mortality Among Persons Entering HIV Care Compared With the General US Population: An Observational Study. *Annals of Internal Medicine*. 2021.
- 204. Curley J, Ssewamala F, Han C-K. Assets and Educational Outcomes: Child Development Accounts (CDAs) for Orphaned Children in Uganda. *Children and youth services review.* 2010;32(11):1585-1590.
- 205. Ismayilova L, Ssewamala F, Mooers E, Nabunya P, Sheshadri S. Imagining the future: Community perceptions of a family-based economic empowerment intervention for AIDS-orphaned adolescents in Uganda. *Children and youth services review.* 2012;34(10):2042-2051.
- 206. Kagotho N, Ssewamala FM. Correlates of depression among caregivers of children affected by HIV/AIDS in Uganda: Findings from the Suubi-Maka Family Study. *AIDS care*. 2012;24(10):1226-1232.
- 207. Ssewamala FM, Neilands TB, Waldfogel J, Ismayilova L. The impact of a comprehensive microfinance intervention on depression levels of AIDS-orphaned children in Uganda. *Journal of Adolescent Health*. 2012;50(4):346-352.
- 208. Witte SS, Aira T, Tsai LC, et al. Efficacy of a savings-led microfinance intervention to reduce sexual risk for HIV among women engaged in sex work: a randomized clinical trial. *American Journal of Public Health*. 2015;105(3):e95-e102.
- 209. Ssewamala FM, Bahar OS, McKay MM, Hoagwood K, Huang K-Y, Pringle B. Strengthening mental health and research training in Sub-Saharan Africa (SMART Africa): Uganda study protocol. *Trials.* 2018;19(1):423.
- 210. Ssewamala FM, Bermudez LG, Neilands TB, et al. Suubi4Her: a study protocol to examine the impact and cost associated with a combination intervention to prevent HIV risk behavior and improve mental health functioning among adolescent girls in Uganda. *BMC public health*. 2018;18(1):693.
- 211. Wang JSH, Ssewamala FM, Neilands TB, et al. Effects of Financial Incentives on Saving Outcomes and Material Well-Being: Evidence From a Randomized Controlled Trial in Uganda. *Journal of Policy Analysis and Management*. 2018;37(3):602-629.
- 212. Uganda AIDS Commission, Ministry of Health, UNAIDS. *HIV and AIDS Uganda country progress report 2016-2017*. Kampala, Uganda2016-2017.
- 213. Chang LW, Grabowski MK, Ssekubugu R, et al. Heterogeneity of the HIV epidemic in agrarian, trading, and fishing communities in Rakai, Uganda: an observational epidemiological study. *The lancet HIV*. 2016;3(8):e388-e396.
- 214. Coates J, Swindale A, Bilinsky P. Household Food Insecurity Access Scale (HFIAS) for measurement of food access: indicator guide: version 3. 2007.





- 215. Radloff LS. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1977;1(3):385-401.
- 216. Beck AT, Steer RA, Pompili M. *BHS, Beck hopelessness scale: manual.* Psychological corporation San Antonio, TX; 1988.
- 217. Coelho GLH, Vilar R, Hanel PHP, Monteiro RP, Ribeiro MGC, Gouveia VV. Optimism scale: Evidence of psychometric validity in two countries and correlations with personality. *Personality and Individual Differences*. 2018;134:245-251.
- 218. Cohen S, Kamarck T, Mermelstein R. Perceived stress scale (PSS). J Health Soc Beh. 1983;24:285.
- 219. Landmark T, Romundstad P, Dale O, Borchgrevink PC, Kaasa S. Estimating the prevalence of chronic pain: validation of recall against longitudinal reporting (the HUNT pain study). *Pain.* 2012;153(7):1368-1373.
- 220. National Institute on Drug Abuse (NIDA). NIDA-Modified Alcohol Smoking and Substance Involvement Screening Test (NM-ASSIST). In.
- 221. Russell DW. UCLA Loneliness Scale (Version 3): Reliability, validity, and factor structure. *Journal of personality assessment.* 1996;66(1):20-40.
- 222. Stark L, Seff I, Hoover A, Gordon R, Ligiero D, Massetti G. Sex and age effects in past-year experiences of violence amongst adolescents in five countries. *PloS one*. 2019;14(7):e0219073-e0219073.
- 223. Chiang LF, Kress H, Sumner SA, Gleckel J, Kawemama P, Gordon RN. Violence Against Children Surveys (VACS): towards a global surveillance system. *Inj Prev.* 2016;22 Suppl 1(Suppl 1):i17-22.
- 224. Zimet GD, Dahlem NW, Zimet SG, Farley GK. The multidimensional scale of perceived social support. *Journal of personality assessment.* 1988;52(1):30-41.
- 225. Moos RH. *Family environment scale manual: Development, applications, research.* Consulting Psychologists Press; 1994.
- 226. Skinner HA, Steinhauer PD, Santa-Barbara J. The family assessment measure. *Canadian Journal of Community Mental Health.* 2009;2(2):91-103.
- 227. Murphy A, Steele M, Dube SR, et al. Adverse Childhood Experiences (ACEs) Questionnaire and Adult Attachment Interview (AAI): Implications for parent child relationships. *Child Abuse & Neglect*. 2014;38(2):224-233.
- 228. Shato T, Nabunya P, Byansi W, et al. Family Economic Empowerment, Family Social Support, and Sexual Risk-Taking Behaviors Among Adolescents Living With HIV in Uganda: The Suubi+Adherence Study. *Journal of Adolescent Health.* 2021.
- 229. Berger BE, Ferrans CE, Lashley FR. Measuring stigma in people with HIV: Psychometric assessment of the HIV stigma scaleH *Research in nursing & health.* 2001;24(6):518-529.
- 230. Wilson IB, Lee Y, Michaud J, Fowler FJ, Jr., Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. *AIDS and behavior*. 2016;20(11):2700-2708.



- 231. Jalali MS, Botticelli M, Hwang RC, Koh HK, McHugh RK. The opioid crisis: a contextual, social-ecological framework. *Health Research Policy and Systems*. 2020;18(1):87.
- 232. PATH. *Life Planning Skills: A Curriculum for Young People in Africa Uganda Version Facilitator's Manual.*Washington, D.C.2003.
- 233. Ssewamala FM, Ismayilova L, McKay M, Sperber E, Bannon W, Alicea S. Gender and the Effects of an Economic Empowerment Program on Attitudes Toward Sexual Risk-Taking Among AIDS-Orphaned Adolescent Youth in Uganda. *Journal of Adolescent Health*. 2010;46(4):372-378.
- 234. Jennings L, Ssewamala FM, Nabunya P. Effect of savings-led economic empowerment on HIV preventive practices among orphaned adolescents in rural Uganda: results from the Suubi-Maka randomized experiment. *AIDS Care.* 2016;28(3):273-282.
- 235. Ssewamala FM, Han C-K, Neilands TB. Asset ownership and health and mental health functioning among AIDS-orphaned adolescents: Findings from a randomized clinical trial in rural Uganda. *Social Science & Medicine*. 2009;69(2):191-198.
- 236. NVIVO 12 [computer program]. QSR International; 2018.
- 237. Lincoln YS, & Guba, E. G. Naturalistic inquiry. Newbury Park, CA: Sage Publications; 1985.
- 238. Strauss A, & Corbin, J. . *Basics of qualitative research: Techniques and procedures for developing grounded theory.* 2nd ed. Thousand Oaks, CA: Sage; 1998.
- 239. Charmaz K. Grounded Theory: Objectivist and Constructivist Methods. Handbook of Qualitative Research. NK Denzin and YS Lincoln. In: Thousand Oaks, Sage Publications; 2000.
- 240. Boyatzis RE. Transforming qualitative information: Thematic analysis and code development. sage; 1998.
- 241. Padgett DK. Qualitative methods in social work research. Vol 36: Sage publications; 2016.
- 242. Creswell JW, Clark VLP. Designing and conducting mixed methods research. Sage publications; 2017.
- 243. Greene JC, Caracelli VJ. Advances in mixed-method evaluation: The challenges and benefits of integrating diverse paradigms. Jossey-Bass; 1997.
- 244. Greene JC, Caracelli VJ, Graham WF. Toward a conceptual framework for mixed-method evaluation designs. *Educational evaluation and policy analysis*. 1989;11(3):255-274.
- 245. Ministry of Health Uganda. Child and Adolescent Mental Health Policy Guidelines. 2017.



